CLINICAL TRIAL: NCT07142161
Title: A Study on the Safety, Preliminary Efficacy, and Cellular Kinetics of Allogeneic CD7-targeted CAR-T Cell Injection in the Treatment of Type 1 Diabetes
Brief Title: A Study on the Safety, Preliminary Efficacy, and Cellular Kinetics of Allo-CD7 CAR-T Cells in T1DM
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD13-02T-AS
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD13-02 (Experimental): CAR T-cell therapy administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphami
  Interventions: Drug: RD13-02 cell infusion

INTERVENTIONS:
Drug: RD13-02 cell infusion — CAR T-cell therapy administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphami

SUMMARY:
This is an open clinical pharmacological translational Research Study, aiming to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of RD13-02 in patients with aT1DM

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes presenting with any of the following conditions:

Impaired hypoglycemia awareness (lack of sufficient autonomic symptoms when plasma glucose is below 54 mg/dL [3 mmol/L]) or other clinically diagnosed neuropathy caused by type 1 diabetes, including but not limited to gastrointestinal autonomic neuropathy Metabolic instability: two or more previous severe hypoglycemic events that required assistance from others, or two or more hospitalizations for ketoacidosis in the past year

* Age ≤ 60 years
* Body weight ≥ 40 kg
* At least one positive islet autoantibody, including glutamic acid decarboxylase autoantibody (GADA), protein tyrosine phosphatase autoantibody (IA-2A), insulin autoantibody (IAA) (only applicable within 2 weeks of insulin treatment), zinc transporter 8 antibody (ZnT8), islet cell autoantibody (ICA), etc.
* MMTT stimulated C-peptide peak > 0.1 nmol/L, or fasting C-peptide > 0.05 nmol/L
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test at screening
* Both male and female subjects must be willing to use contraception from the time of signing the informed consent form until 12 months after cell infusion
* The subject or their legal guardian voluntarily participates in this study and is able to sign the informed consent form

Exclusion Criteria:

* If any of the following criteria are met, the subject will be excluded from the study.

Type 2 diabetes, or diabetes mellitus from pregnancy, single-gene mutation, pancreatic injury, or other secondary causes (e.g., Cushing's syndrome, thyroid dysfunction, or acromegaly)

* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 x ULN, or total bilirubin ≥ 1.5 x ULN
* Severe heart disease, with any of the following:
* Myocardial infarction within 1 year before enrollment
* Signs or symptoms of heart failure of NYHA Class ≥ 3 within 1 year before enrollment
* Left ventricular ejection fraction (LVEF) < 50% at screening
* QTcF > 450 msec (males) or > 470 msec (females), based on the QTcF value from a single ECG or the average of three repeated ECGs taken more than 3 minutes apart (QT interval corrected by Fridericia's formula)
* Severe concurrent diabetic nephropathy, with an estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2
* Currently undergoing or expected to require renal replacement therapy during the study
* At screening, a subject tests positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B e-antigen (HBeAg); a subject tests positive for hepatitis B e-antibody (HBeAb) with a peripheral blood HBV DNA level above the upper limit of normal; a subject tests positive for hepatitis C virus (HCV) antibody; a subject tests positive for human immunodeficiency virus (HIV) antibody; a subject tests positive for syphilis antibody; a subject tests positive for EBER or has an EBV viral load greater than the upper limit of normal
* Participated in another clinical study within 3 months prior to enrollment
* Received a live attenuated vaccine within 4 weeks prior to enrollment
* The investigator considers the patient to have latent T1DM, including latent autoimmune diabetes in adults (LADA) and latent autoimmune diabetes in the young (LADY)
* The investigator believes there are other reasons that make the subject unsuitable for this clinical study

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicity (DLT) of RD13-02 in patients with type 1 diabetes, as well as the incidence of adverse events (AE), serious adverse events (SAE), and adverse events of special interest (AESI) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Bioheng, Nanjing, China

IPD SHARING:
Plan to Share IPD: No